CLINICAL TRIAL: NCT05226416
Title: Analysis of Health Status of Сomorbid Adult Patients With COVID-19 Hospitalised in Fourth Wave of SARS-CoV-2 Infection (ACTIV4)
Brief Title: Analysis of Health Status of Сomorbid Adult Patients With COVID-19 Hospitalised in Fourth Wave of SARS-CoV-2 Infection
Acronym: ACTIV4
Status: Completed | Type: Observational
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Principal Investigator, Tamara Kriukova, Head of Organizational Committee, Eurasian Association of Therapists
Other Study IDs: ACTIV4
Record Dates: First submitted 2022-02-01; First posted 2022-02-07 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; Chronic Heart Failure; Diabetes Mellitus; Chronic Kidney Diseases; Ischemic Heart Disease; Arrythmia; Hypertensive Heart Disease; Overweight and Obesity; Oncology; Ischemic Stroke; Myocardial Infarction; Atrial Fibrillation; DVT; Stroke; Copd; Asthma; Pulmonary Embolism; Anemia; Myocarditis
Keywords: covid-19; ACTIV; Chronic Heart Failure; Ischemic Heart Disease; Hypertensive Heart Disease; Chronic Kidney Diseases; Atrial Fibrillation; Myocarditis
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Renal Insufficiency, Chronic; Myocardial Ischemia; Arrhythmias, Cardiac; Overweight; Obesity; Neoplasms; Ischemic Stroke; Myocardial Infarction; Atrial Fibrillation; Stroke; Pulmonary Disease, Chronic Obstructive; Asthma; Pulmonary Embolism; Anemia; Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Depersonalized multi-centered registry initiated to analyze dynamics of non-infectious diseases after SARS-CoV-2 infection in population of Eurasian adult patients.

DETAILED DESCRIPTION:
Assessment of hospital course and health status during 3, 6, 12 months after discharge in COVID-19 patients in cohorts with comorbidities and without comorbidities. Evaluation of comorbidity impact to severity of novel coronavirus disease and comorbidity impact to demand for medical care.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed COVID-19

Exclusion Criteria:

* Age under 18 years.
* Refusal to be involved in study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anonymized male and female patients over 18 years hospitalized with COVID-19 during the fourth wave of novel coronavirus disease.
Sampling Method: Probability Sample
Enrollment: 3554 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
death for any cause | From date of hospitalization until the date of first documented date of death from any cause, assessed up to 12 months
  rate of lethal outcomes
hospitalization for any cause | 12 months after discharge
  rate of hospitalization for any cause

SECONDARY OUTCOMES:
onset of any disease diagnosed 1 year after discharge | 1 year after discharge
  rate of patients with onset of any disease diagnosed 1 year after discharge
rate of demand for medical care | 1 year after discharge
  number of patients seeking for health care after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Arutyunov, MD, PhD, Principal Investigator — Eurasian Association of Therapists
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No